CLINICAL TRIAL: NCT04607460
Title: Biofeedback EMG Alternative Therapy for Chronic Low Back Pain and Chronic Cancer Pain (BEAT-Pain): A Pilot Efficacy Study
Brief Title: EMG Biofeedback Treatment for Chronic Low Back Pain, Cancer Pain and Migraines
Acronym: BEAT-Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Asimina Lazaridou, PhD, Instructor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020P003158
Record Dates: First submitted 2020-10-06; First posted 2020-10-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Chronic Low-back Pain; Mastectomy; Lumpectomy; Migraine
Keywords: EMG-Biofeedback; Chronic low-back pain; Mastectomy; Lumpectomy; Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (6):
- EMG-Biofeedback for Lower Back Pain (Experimental): Participants will receive a JOGO Digital Therapeutics EMG Biofeedback device and a software installed on a tablet or smart phone. During the 8 weekly sessions participants will be instructed on how to use the device by a trained biofeedback instructor.
  Interventions: Device: JOGO Digital Therapeutics EMG Biofeedback for Lower Back Pain
- Treatment as usual (Lower Back Pain) (No Intervention): Participants in this group will receive no active treatment.
- EMG-Biofeedback for Persistent Post-Mastectomy Pain (Experimental): Participants will receive a JOGO Digital Therapeutics EMG Biofeedback device and a software installed on a tablet or smart phone. During the 4 weekly sessions participants will be instructed on how to use the device by a trained biofeedback instructor ahead of their mastectomy.
  Interventions: Device: JOGO Digital Therapeutics EMG Biofeedback for Persistent Post Mastectomy Pain
- Treatment as usual (Persistent Post-Mastectomy Pain) (No Intervention): Participants in this group will receive no active treatment.
- EMG-Biofeedback for Migraine (Experimental): Participants will receive a JOGO Digital Therapeutics EMG Biofeedback device and a software installed on a tablet or smart phone. During the 6 weekly sessions participants will be instructed on how to use the device by a trained biofeedback instructor.
  Interventions: Device: JOGO Digital Therapeutics EMG Biofeedback for Migraine
- Treatment as usual (Migraine) (No Intervention): Participants in this group will receive no active treatment.

INTERVENTIONS:
Device: JOGO Digital Therapeutics EMG Biofeedback for Lower Back Pain — Use of the JOGO Digital Therapeutics EMG Biofeedback device for 8 weeks with specific exercises to target low back pain.
  Arms: EMG-Biofeedback for Lower Back Pain
Device: JOGO Digital Therapeutics EMG Biofeedback for Persistent Post Mastectomy Pain — Use of the JOGO Digital Therapeutics EMG Biofeedback device for 4 weeks with specific exercises to mitigate persistent post mastectomy pain ahead of the surgery.
  Arms: EMG-Biofeedback for Persistent Post-Mastectomy Pain
Device: JOGO Digital Therapeutics EMG Biofeedback for Migraine — Use of the JOGO Digital Therapeutics EMG Biofeedback device for 6 weeks with specific exercises to target migraine pain.
  Arms: EMG-Biofeedback for Migraine

SUMMARY:
The purpose of this pilot efficacy study is to examine the effects of EMG-biofeedback (EMG-BF) on pain-related outcomes in Chronic Low Back Pain (CLBP) patients, Recent mastectomy and lumpectomy patients, and patients with episodic migraine.

EMG-BF facilitates neuromuscular retraining and muscle relaxation by using audio and visual stimuli using an EMG surface electrode-based biosensor and a software installed on a tablet or smart phone.

For this pilot efficacy study, we will recruit 125 patients with chronic low back pain, 125 patients who are expected to undergo mastectomy and 80 patients with episodic migraine. Participants will be randomly assigned to either the JOGO Digital Therapeutics EMG Biofeedback device or treatment as usual control group.

Patients assigned to the intervention group will be asked to complete self-report questionnaires assessing demographics, pain intensity, negative affect, physical function, pain catastrophizing and sleep, will undergo QST and will be asked to wear Actiwatches to keep track of health behaviors, prior to and after completing the intervention. The intervention consists of weekly sessions during which participants will be instructed on how to use the device by a trained biofeedback instructor.

Patients in the control group will undergo sensory testing procedures at baseline and after treatment period but will receive no active treatment.

The aims of this study are to examine the impact of EMG-BF on pain and QST and the impact of EMG-BF on psychosocial function. We hypothesize that patients that will undergo the EMG-BF will demonstrate reductions in pain, physical functioning, sleep, pain catastrophizing, anxiety and depression.

DETAILED DESCRIPTION:
Biofeedback can be described as "operant conditioning of physiological activity", by which "the patient learns to self-regulate his or her physiological processes with the help of feedback information", and can comprise different sites, modalities, and procedures. Biofeedback instruments measure physiological activity such as brainwaves, heart function, breathing, muscle activity, and skin temperature and rapidly and accurately provide feedback information to the user. There are various aims biofeedback can target, e.g., developing more awareness or control for physiological processes and thus, consciously reducing muscle tension. Previous research has shown findings of higher baseline muscle activation and abnormal EMG as a response to stress in chronic back pain patients.

Studies using biofeedback for the treatment of chronic back pain have shown inconsistent results and it is difficult to draw conclusions based on previous studies due to variability in sample size and characteristics, biofeedback modality, treatment conditions, and control groups. Thus, the effectiveness of biofeedback in reducing the symptomatology of back pain patients remains unclear. The investigators therefore are planning to conduct this pilot efficacy study, to examine the effects of EMG-biofeedback (EMG-BF) on pain-related outcomes in a cohort of Chronic Low Back Pain (CLBP) patients.

This randomized clinical trial has two study arms. Participants in the first arm will receive the experimental condition (EMG-Bf) and those in the second will continue their usual care and serve as a control group. Both groups will be asked to complete self-report questionnaires before their first visit and after the last visit at 8 weeks. Further, both groups will undergo Quantitative Sensory Testing (QST) before their first visit and after the last visit at 8 weeks. The specific aims of this study are to examine the impact of EMG-BF on pain intensity and sensitivity and on physical functioning, sleep, pain catastrophizing, anxiety and depression. We will not modify pain medication regimens in any of the trial arms and no pain medication prescriptions will be issued by the research team at any time.

Chronic Lower Back Pain

Experimental Condition:

This study will include 2 in-person office visits separated by 8 virtual therapy sessions. During the in-person visits, participants will undergo sensory testing procedures described below. On visit 1 a member of the research staff will train patients on the basic functionality of the EMG-BF device. Virtual sessions 1-8 will be held via Partners Healthcare Secure Zoom. During these, participants will receive guided EMG biofeedback intervention with a therapist and will be instructed to use the device at home.

Home practice will be monitored via electronic practice logs recorded on REDcap. Patients will be trained to relax their muscles under the guidance of a doctorate level therapist by monitoring progress through virtual feedback in the form of graph.

Treatment as Usual: Patients in this group will undergo sensory testing procedures described below at baseline and after 8 weeks but will receive no active treatment.

Chronic Cancer Pain

Experimental Condition:

This study will include 2 in-person office visits separated by 2 weekly virtual therapy sessions before and 2 virtual therapy sessions after their scheduled mastectomy as well as a period of 3 months after their procedure. During the in-person visits, participants will undergo sensory testing procedures described below. On visit 1 a member of the research staff will train patients on the basic functionality of the EMG-BF device. Virtual sessions 1 and 2 will be held via Partners Healthcare Secure Zoom ahead of their scheduled mastectomy and sessions 3 and 4 will be held after. During these, participants will receive guided EMG biofeedback intervention with a therapist and will be instructed to use the device at home.

Home practice will be monitored via electronic practice logs recorded on REDcap. Patients will be trained to relax their muscles under the guidance of a doctorate level therapist by monitoring progress through virtual feedback in the form of graph.

Treatment as Usual: Patients in this group will undergo sensory testing procedures described below at baseline and 3 months after their mastectomy but will receive no active treatment.

Migraine Pain

Experimental Condition:

This study will include 2 in-person office visits separated by 6 virtual therapy sessions. During the in-person visits, participants will undergo sensory testing procedures described below. On visit 1 a member of the research staff will train patients on the basic functionality of the EMG-BF device. Virtual sessions 1-6 will be held via Partners Healthcare Secure Zoom. During these, participants will receive guided EMG biofeedback intervention with a therapist and will be instructed to use the device at home.

Home practice will be monitored via electronic practice logs recorded on REDcap. Patients will be trained to relax their muscles under the guidance of a doctorate level therapist by monitoring progress through virtual feedback in the form of graph.

Treatment as Usual: Patients in this group will undergo sensory testing procedures described below at baseline and after 6 weeks but will receive no active treatment.

1) EMG-Biofeedback EMG-BF facilitates neuromuscular retraining and muscle relaxation by using audio and visual stimuli using an EMG surface electrode-based biosensor and a software installed on a tablet or smart phone. During the weekly sessions participants will be instructed on how to use the device by a trained biofeedback instructor. Further, in each session participants will have the opportunity to discuss possible difficulties/obstacles/progress using the device. Each session will additionally include relaxation techniques (such as Progressive Muscle Relaxation). Sessions are estimated to last 40-45 minutes.

Standardized Quantitative Sensory Testing (QST) QST is a non-invasive method for measuring pain sensitivity and pain modulation. Our QST testing protocol will measure mechanical pain sensitivity (pain threshold). This protocol has been used in various studies the investigators have conducted in the past. During the psychophysical testing procedures, participants will be informed that they may terminate the procedure at any time. The intensity of pain stimulation will be determined for each subject individually to minimize potential for tissue damage. The methods used have been thoroughly tested and validated for the study of experimental pain. All subjects will be examined during the study to document the presence or absence of tissue injury at the sites of noxious stimulation. If there is any evidence that the protocol causes more than minor, reversible bruising or sensitization, the protocol will be amended to decrease the frequency and/or intensity of the noxious stimuli. Outcome monitoring and adverse events will all be reported through appropriate channels of the Human Studies Committee.

ELIGIBILITY:
Low Back Pain

Inclusion Criteria:

* Age 18-65 years old;
* Chronic Low Back Pain as seen on medical history for at least 6 months but no longer than 10 years;
* A minimum score of >3 on pain visual analog scale (VAS) at the start of experimental sessions;
* are able to speak and understand English, and (6) have access to a computer or tablet at home and have an email address.

Exclusion Criteria:

* Lower back surgery within previous twelve (12) months;
* Comorbid chronic pain condition that is rated by the subject as more painful than CLBP
* Pain condition requiring urgent surgery;
* Females who are pregnant;
* Subjects with a severe visual or hearing impairment;
* Evidence of non-mechanical contributing cause for lower back pain e.g. neoplasm, infection, fracture, inflammatory disorder incl. acute osteomyelitis or acute bone disease;
* Subjects currently under active cancer treatment (chemo, infusion, ongoing radiation);
* Implanted medical device (spinal cord stimulator, intrathecal pump or peripheral nerve stimulator);
* Medical condition known to influence QST or participation in the EMG intervention
* (e.g. HIV, peripheral neuropathy, Raynaud's syndrome);
* Present or past serious psychiatric condition (e.g. Schizophrenia, delusional disorder,
* psychotic disorder, or dissociative disorder) or any psychiatric condition that required hospitalization the past year and that would be judged to interfere with study participation.
* Active addiction disorder, such as cocaine or IV heroin use, that would interfere with
* study participation,
* Diagnosis of mild cognitive impairment or dementia
* Significant medical abnormalities or conditions that in the opinion of the Practitioner
* would interfere either with the ability to complete the study or the evaluation of the investigational device's safety and efficacy.
* Recent history of a significant medical-surgical intervention that in the judgment of the
* Practitioner would interfere either with the ability to complete the study or the evaluation of the investigative device's safety and efficacy.
* Known allergic skin reaction to tapes and plasters.
* Subject who is currently enrolled in an investigational drug or device study.

Chronic Cancer Pain

Inclusion criteria:

* Female
* Aged 18-65 years old
* Recent bodily pain complaints with a minimum score of >1 on pain visual analog scale (VAS) at the start of experimental sessions;
* Scheduled for breast biopsy
* Willingness to undergo psychophysical and psychosocial testing
* Willingness to participate in long-term follow-up are able to speak and understand English, and (8) have access to a computer or tablet at home and have an email address.

Exclusion criteria:

* Pregnant
* Present or past serious psychiatric condition (e.g. Schizophrenia, delusional disorder, psychotic disorder, or dissociative disorder) or any psychiatric condition that required hospitalization the past year and that would be judged to interfere with study participation.
* Pain condition requiring urgent surgery;
* Subjects with a severe visual or hearing impairment;
* Implanted medical device (spinal cord stimulator, intrathecal pump or peripheral nerve stimulator);
* Medical condition known to influence QST or participation in the EMG intervention (e.g. HIV, peripheral neuropathy, Raynaud's syndrome);
* Active addiction disorder, such as cocaine or IV heroin use, that would interfere with study participation,
* Diagnosis of mild cognitive impairment or dementia
* Significant medical abnormalities or conditions that in the opinion of the Practitioner would interfere either with the ability to complete the study or the evaluation of the investigational device's safety and efficacy.
* Recent history of a significant medical-surgical intervention that in the judgment of the Practitioner would interfere either with the ability to complete the study or the evaluation of the investigative device's safety and efficacy.
* Known allergic skin reaction to tapes and plasters.
* Subject who is currently enrolled in an investigational drug or device study.

Migraine Pain

Inclusion Criteria:

* Women ages 18-65
* Diagnosis of episodic migraine (with or without aura) (International Classification of Headache Disorders-II)(15)
* 4-14 days with migraine in the last month
* No change in the type of prophylactic and psychiatric medication used within the last 3 months
* Greater than one year of migraines (self-reported)
* Agreeable to participate, commit to all study procedures, and to be randomized to either group
* Fluent in English (required to complete self-report instruments)

Exclusion Criteria:

* Any unstable medical (e.g. neurodegenerative conditions) or psychiatric conditions (e.g. psychosis) requiring immediate treatment or that could lead to difficulty complying with the protocol
* Active suicidal ideation (assessed by the clinician during initial screening)
* Moderate or severe level of depression (exclude if score on PHQ-2 is greater than or equal to 3)
* Psychiatric hospitalization within the past year (self-reported)
* Comorbid acute or chronic pain condition that is rated by the subject as more painful than migraine
* Begins new migraine treatment during the study period
* Inability to complete study visits
* Medical condition known to influence QST or participation in the EMG intervention (e.g. HIV, peripheral neuropathy, Raynaud's syndrome);
* Active addiction disorder, such as cocaine or IV heroin use, that would interfere with study participation,
* Significant medical abnormalities or conditions that in the opinion of the Practitioner would interfere either with the ability to complete the study or the evaluation of the investigational device's safety and efficacy.
* Recent history of a significant medical-surgical intervention that in the judgment of the Practitioner would interfere either with the ability to complete the study or the evaluation of the investigative device's safety and efficacy.
* Known allergic skin reaction to tapes and plasters.
* Subject who is currently enrolled in an investigational drug or device study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Pain intensity after treatment period | Through study completion, an average of 6 months
  will be assessed using the 0-10-point Numerical Rating Scale (NRS) from the Brief Pain Inventory (BPI) assessing pain intensity and pain interference.

SECONDARY OUTCOMES:
Negative affect (anxiety, depression) | Through study completion, an average of 6 months
  will be assessed by the Hospital Anxiety and Depression Scale. Score range 0 and 21 for either anxiety or depression, where higher scores indicate higher anxiety or depression respectively
Physical function | Through study completion, an average of 6 months
  will be measured using the validated Oswestry Disability Index (ODI). Score range 0-100, where higher scores indicate greater disability/functional impairment
Pain catastrophizing | Through study completion, an average of 6 months
  will be assessed with the Pain Catastrophizing Scale (PCS). Score range 0-52, where higher scores indicate greater pain catastrophizing.
Sleep Quality | Through study completion, an average of 6 months
  will be assessed using the Pittsburgh Sleep Quality Index (PSQI). The score can range between 0-21, the higher the score, the worse the sleep quality.
Pain sensitivity in kPa (pain threshold) | Through study completion, an average of 6 months
  Pressure pain threshold will be assessed using a digital pressure algometer. Unit of Measure: lbf
Pain sensitivity in mmHg (pain threshold) | Through study completion, an average of 6 months
  Pressure pain threshold will be assessed using a Hokanson rapid cuff inflator. Unit of Measure: mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Asimina Lazaridou, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD

REFERENCES:
- [Background] Schwartz MS, Andrasik F. Biofeedback : a practitioner's guide. Fourth edition. ed. New York: The Guilford Press; 2016.
- [Background] Sielski R, Glombiewski JA. Biofeedback as a psychological treatment option for chronic back pain. Pain Manag. 2017 Mar;7(2):75-79. doi: 10.2217/pmt-2016-0040. Epub 2016 Nov 4. No abstract available. PMID 27809657
- [Background] Jacobs JV, Henry SM, Jones SL, Hitt JR, Bunn JY. A history of low back pain associates with altered electromyographic activation patterns in response to perturbations of standing balance. J Neurophysiol. 2011 Nov;106(5):2506-14. doi: 10.1152/jn.00296.2011. Epub 2011 Jul 27. PMID 21795622
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Snaith RP. The hospital anxiety and depression scale. Br J Gen Pract. 1990 Jul;40(336):305. No abstract available. PMID 2081070
- [Background] Sullivan MJ, Thorn B, Haythornthwaite JA, Keefe F, Martin M, Bradley LA, Lefebvre JC. Theoretical perspectives on the relation between catastrophizing and pain. Clin J Pain. 2001 Mar;17(1):52-64. doi: 10.1097/00002508-200103000-00008. PMID 11289089
- [Background] Smyth C. The Pittsburgh Sleep Quality Index (PSQI). Director. 2000 Winter;8(1):28-9. No abstract available. PMID 11081020
- [Background] Katz NP, Paillard FC, Edwards RR. Review of the performance of quantitative sensory testing methods to detect hyperalgesia in chronic pain patients on long-term opioids. Anesthesiology. 2015 Mar;122(3):677-85. doi: 10.1097/ALN.0000000000000530. PMID 25437498
- [Background] Wasan AD, Alter BJ, Edwards RR, Argoff CE, Sehgal N, Walk D, Moeller-Bertram T, Wallace MS, Backonja M. Test-Retest and Inter-Examiner Reliability of a Novel Bedside Quantitative Sensory Testing Battery in Postherpetic Neuralgia Patients. J Pain. 2020 Jul-Aug;21(7-8):858-868. doi: 10.1016/j.jpain.2019.11.013. Epub 2019 Dec 11. PMID 31837446
- [Background] Jamison RN, Jurcik DC, Edwards RR, Huang CC, Ross EL. A Pilot Comparison of a Smartphone App With or Without 2-Way Messaging Among Chronic Pain Patients: Who Benefits From a Pain App? Clin J Pain. 2017 Aug;33(8):676-686. doi: 10.1097/AJP.0000000000000455. PMID 27898460
- [Background] Jamison RN, Xu X, Wan L, Edwards RR, Ross EL. Determining Pain Catastrophizing From Daily Pain App Assessment Data: Role of Computer-Based Classification. J Pain. 2019 Mar;20(3):278-287. doi: 10.1016/j.jpain.2018.09.005. Epub 2018 Sep 29. PMID 30273687
- [Background] Lazaridou A, Paschali M, Vilsmark ES, Edwards RR. Biofeedback EMG alternative therapy for chronic low back pain: Study protocol of a pilot randomized controlled trial. Contemp Clin Trials. 2022 Oct;121:106888. doi: 10.1016/j.cct.2022.106888. Epub 2022 Aug 18. PMID 35988661
- [Result] Lazaridou A, Paschali M, Vilsmark ES, Sadora J, Burton D, Bashara A, Edwards RR. Biofeedback EMG alternative therapy for chronic low back pain (the BEAT-pain study). Digit Health. 2023 Feb 7;9:20552076231154386. doi: 10.1177/20552076231154386. eCollection 2023 Jan-Dec. PMID 36776410
- [Result] Sadora J, Vilsmark E, Bashara A, Burton D, Paschali M, Pester B, Curiel M, Edwards R, Lazaridou A. Electromyography-biofeedback for chronic low back pain: A qualitative cohort study. Complement Ther Med. 2023 May;73:102922. doi: 10.1016/j.ctim.2023.102922. Epub 2023 Jan 28. PMID 36716896